CLINICAL TRIAL: NCT05662865
Title: Low-CArbohydrate Diet and SGLT2-INhibitOr to Achieve Moderate Ketosis in Healthy Volunteers (CASINO)
Brief Title: Low-CArbohydrate Diet and SGLT2-INhibitOr to Achieve Moderate Ketosis in Healthy Volunteers
Acronym: CASINO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1921572
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Ketones, Metabolism
MeSH Terms: conditions — Ketosis | interventions — Sodium-Glucose Transporter 2 Inhibitors; ertugliflozin; Control Groups

STUDY DESIGN:
Intervention Model Description: Proof-of-concept, single-group, study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single, Experimental Group (Experimental): SGLT2i + adaptive study diet of progressive dietary carbohydrate reduction
  Interventions: Drug: SGLT2 inhibitor; Other: Controlled, Adaptive Study Diet

INTERVENTIONS:
Drug: SGLT2 inhibitor — SGTL2i (15 mg) once daily
  Other Names: ertugliflozin
Other: Controlled, Adaptive Study Diet — An adaptive study diet combined with SGLT2i, which consists of four sequential, 7-day long phases in which dietary carbohydrates are gradually reduced (50% carbs, 30% carbs, 20% carbs, and 10% carbs) based on safety and tolerability to achieve moderate ketosis. All diet phases are isocaloric. All meals are provided on an inpatient unit.

SUMMARY:
The purpose of this study is to help us better understand how plasma ketones respond to a low-carb diet when combined with an SGLT2 inhibitor.

DETAILED DESCRIPTION:
We will combine an SGLT2i with an adaptive study diet that gradually reduces dietary carbohydrates to safely achieve moderate ketosis in healthy adult volunteers.

ELIGIBILITY:
Inclusion criteria:

* M/F
* Age 18-60 years
* Weight stable (+/- 3 kg over past 6 months)
* Body mass index (BMI): 21-35 kg/m2
* Otherwise healthy, as determined by medical history and laboratory tests
* Understands the procedures and agrees to participate by giving written informed consent
* Willing and able to comply with scheduled visits, laboratory tests, and other study procedures

Exclusion criteria:

Acute or chronic medical conditions or medication that would contraindicate the participation in the research testing or could potentially affect metabolic function including, but not limited to:

1. History or presence of cardiovascular disease (unstable angina, myocardial infarction or coronary revascularization within 6 months, presence of cardiac pacemaker, implanted cardiac defibrillator)
2. Diagnosis of type 1 or type 2 diabetes mellitus, or prior diabetic ketoacidosis
3. Blood pressure > 140/90 mm Hg
4. Bleeding and clotting disorders
5. Acute or chronic infection (such as TB, HIV or Hepatitis)
6. Renal insufficiency (eGFR<60), nephritis, or chronic kidney disease
7. Thyroid dysfunction (suppressed TSH, elevated TSH <10 µIU/ml if symptomatic or elevated TSH >10 µIU/ml if asymptomatic)
8. Liver disease (liver function tests > 2 x normal; including NASH/NAFLD)
9. Gastrointestinal disorders (including inflammatory bowel disease or malabsorption, swallowing disorders, suspected or known strictures, fistulas or physiological/mechanical GI obstruction, history of gastrointestinal surgery, Crohn's disease or diverticulitis)
10. Past or present history of eating disorder (including binge eating)
11. Past or present history of psychiatric disease, including major depressive illness or bipolar disorder, as well as claustrophobia since part of the protocol will involve being confined to a small room for whole-body indirect calorimetry
12. Unwilling or unable to eat the foods provided in the study diet
13. A positive urine drug test for illicit drugs.
14. Any malignancy not considered cured, except basal cell carcinoma and squamous cell carcinoma of the skin (a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years)
15. Pregnant or nursing females or females less than 6 months postpartum from the scheduled date of collection
16. Regular smoking or regular nicotine use of any kind including chewing tobacco, snuff and vaping
17. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study days.
18. History of regular alcohol consumption exceeding 7 drinks/week for female participants or 14 drinks/week for male participants (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
19. Donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
20. Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women)

Excluded medications include, but are not limited to:

1. Any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
2. Anti-diabetic agents
3. Recent change to medication and/or dosing in the past 3 months
4. Blood thinner prescription medication
5. Chronic use of aspirin or other non-steroidal anti-inflammatory drugs, including COX-2 inhibitors (a single aspirin daily if prescribed for cardioprotection will be allowed as will occasional use of aspirin and other non-steroidal drugs, provided that they are used for < 3 consecutive days and not during the period of metabolic testing)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fasting ketones | 28 days
  To determine if the primary study objective was achieved (e.g. SGLT2i combined with dietary carbohydrate restriction achieves moderate ketosis, safely and tolerably, in healthy, non-diabetic adults), we will use a binary decision (yes/no) for each participant, based on fasting capillary ketones.

SECONDARY OUTCOMES:
24h AUC plasma ketones | 28 days
  The secondary objective of this study is to analyze changes in fasting and 24h AUC of plasma ketones (BHB and AcAc) between SGLT2i + standard-carb diet versus SGLT2i + low-carb/adaptive diet using within-subject repeated measures analysis of variance. A p-value less than 0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Erickson, PhD, Principal Investigator — AdventHealth Translational Research Institute
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AdventHealth Translational Research Institute, Orlando, FL — https://www.adventhealthresearchinstitute.com/research/translational-research